CLINICAL TRIAL: NCT01345656
Title: A Randomized, Double-blind, Multi-center Study to Assess Safety and Tolerability of Different Oral Doses of BAY94-8862 in Subjects With Stable Chronic Heart Failure With Left Ventricular Systolic Dysfunction and Mild (Part A) or Moderate (Part B) Chronic Kidney Disease Versus Placebo (Part A) or Versus Placebo and Spironolactone (Part B)
Brief Title: BAY94-8862 Dose Finding Trial in Subjects With Chronic Heart Failure and Mild (Part A) or Moderate (Part B) Chronic Kidney Disease
Acronym: ARTS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14563; 2011-000301-45 (EudraCT Number)
Record Dates: First submitted 2011-04-29; First posted 2011-05-02 (Estimated); Last update posted 2022-02-10 (Actual); Status verified 2022-01

CONDITIONS: Heart Failure
Keywords: Chronic Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — finerenone; Spironolactone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Arm 1 (Experimental)
  Interventions: Drug: BAY94-8862
- Arm 2 (Experimental)
  Interventions: Drug: BAY94-8862
- Arm 3 (Experimental)
  Interventions: Drug: BAY94-8862
- Arm 4 (Experimental)
  Interventions: Drug: BAY94-8862
- Arm 5 (Placebo Comparator)
  Interventions: Drug: Placebo
- Arm 6 (Active Comparator)
  Interventions: Drug: Spironolactone

INTERVENTIONS:
Drug: BAY94-8862 — Two 1.25 mg BAY94-8862 and 2 placebo tablets for duration of 4 weeks
  Arms: Arm 1
Drug: BAY94-8862 — Four 1.25 mg BAY94-8862 tablets for duration of 4 weeks
  Arms: Arm 2
Drug: BAY94-8862 — One 10 mg BAY94-8862 tablet for duration of 4 weeks
  Arms: Arm 3
Drug: BAY94-8862 — Part B only: Four 1.25 mg BAY94-8862 tablets in the morning and four tablets in the evening for duration of 4 weeks
  Arms: Arm 4
Drug: Placebo — Placebo tablets for duration of 4 weeks
  Arms: Arm 5
Drug: Spironolactone — Part B only: 25 mg spironolactone once daily with up-titration to 50 mg once daily starting at day 15, if serum potassium is less or equal to 4.8 mmol/L, for duration of 4 weeks
  Arms: Arm 6

SUMMARY:
A placebo (Part A) and placebo and active comparator controlled (Part B), double-blind and randomized study to assess safety and tolerability of a new drug (BAY94-8862) given orally

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18 years and older or postmenopausal women aged 55 years and older or women aged 18 years and older without childbearing potential based on surgical treatment such as bilateral tubal ligation, bilateral ovarectomy, or hysterectomy
* Clinical diagnosis of CHF (chronic heart failure), either ischemic or non-ischemic, NYHA (New York Heart Association) class II - III, treated with evidenced-based therapy for CHF, e.g. beta-blockers and ACE (angiotensin-converting enzyme) inhibitors or ARB (angiotensin receptor blocker) as well as diuretics, unless contraindicated or not tolerated
* Known kidney damage for >/= 3 months, as defined by structural or functional abnormalities of the kidney, and

  * Part A: 60 mL/min/1.73 m*2 </= eGFR (estimated Glomerular Filtration Rate) < 90 mL/min/1.73 m*2 (MDRD, Modification of Diet in Renal Disease) at the screening visit
  * Part B: 30 mL/min/1.73 m*2 </= eGFR <= 60 mL/min/1.73 m*2 (MDRD) at the screening visit
* Serum potassium </= 4.8 mmol/L at the screening visit
* Systolic blood pressure >/= 90 mmHg without signs or symptoms of hypotension at the screening visit

Exclusion Criteria:

* Known hypersensitivity to the study drug (active substance or excipients) or spironolactone and respective excipients (Part B only)
* Subjects with anuria, acute renal failure, or Addison's disease
* Acute coronary syndrome or unstable coronary artery disease within 30 days prior to randomization
* Valvular heart disease requiring surgical intervention during the course of the study
* History of hospitalization for hyperkalemia or acute renal failure induced by previous aldosterone antagonist treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 457 (Actual)
Dates: Start 2011-05-09 (Actual); Primary Completion 2012-05-30 (Actual); Study Completion 2012-07-16 (Actual)

PRIMARY OUTCOMES:
Change of serum potassium | 4 weeks

SECONDARY OUTCOMES:
Change in serum magnesium | Day 8, Day 15, Day 22, Day 29
Change in blood pressure | Day 8, Day 15, Day 22, Day 29
Change in heart rate | Day 8, Day 15, Day 22, Day 29

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (47):
- Austria (3):
  - Graz, Styria
  - Linz, Upper Austria
  - Vienna
- Belgium (3):
  - Brasschaat
  - Bruxelles - Brussel
  - Roeselare
- Czechia (3):
  - Brno
  - Liberec
  - Prague
- Denmark (11):
  - Copenhagen Ø
  - Esbjerg
  - Frederiksberg
  - Hellerup
  - Herlev
  - Hvidovre
  - København NV
  - Køge
  - Odense
  - Svendborg
  - Viborg
- Finland (3):
  - Helsinki
  - Jyväskylä
  - Turku
- Germany (7):
  - Frankfurt am Main, Hesse
  - Cologne, North Rhine-Westphalia
  - Dresden, Saxony
  - Wermsdorf, Saxony
  - Wedel, Schleswig-Holstein
  - Erfurt, Thuringia
  - Berlin
- Israel (7):
  - Afula
  - Ashkelon
  - Hadera
  - Petah Tikva
  - Rehovot
  - Safed
  - Tel Aviv
- Norway (2):
  - Oslo
  - Stavanger
- Poland (5):
  - Krakow
  - Piotrkow Trybunalski
  - Szczecin
  - Warsaw
  - Wroclaw
- Sweden (3):
  - Kristianstad
  - Lund
  - Stockholm

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- [Result] Pitt B, Filippatos G, Gheorghiade M, Kober L, Krum H, Ponikowski P, Nowack C, Kolkhof P, Kim SY, Zannad F. Rationale and design of ARTS: a randomized, double-blind study of BAY 94-8862 in patients with chronic heart failure and mild or moderate chronic kidney disease. Eur J Heart Fail. 2012 Jun;14(6):668-75. doi: 10.1093/eurjhf/hfs061. Epub 2012 May 4. PMID 22562554
- [Result] Pitt B, Kober L, Ponikowski P, Gheorghiade M, Filippatos G, Krum H, Nowack C, Kolkhof P, Kim SY, Zannad F. Safety and tolerability of the novel non-steroidal mineralocorticoid receptor antagonist BAY 94-8862 in patients with chronic heart failure and mild or moderate chronic kidney disease: a randomized, double-blind trial. Eur Heart J. 2013 Aug;34(31):2453-63. doi: 10.1093/eurheartj/eht187. Epub 2013 May 27. PMID 23713082
- [Derived] Ostrominski JW, Filippatos G, Claggett BL, Miao ZM, Desai AS, Jhund PS, Henderson A, Rohwedder K, Brinker MD, Scalise A, Schloemer P, Lam CSP, Senni M, Shah SJ, Voors AA, Zannad F, Rossing P, Ruilope LM, Anker SD, Pitt B, Agarwal R, McMurray JJV, Solomon SD, Vaduganathan M. Effect of Finerenone on Morbidity and Mortality in CKD. J Am Soc Nephrol. 2025 Sep 12. doi: 10.1681/ASN.0000000823. Online ahead of print. No abstract available. PMID 40938666
- [Derived] Chung EY, Ruospo M, Natale P, Bolignano D, Navaneethan SD, Palmer SC, Strippoli GF. Aldosterone antagonists in addition to renin angiotensin system antagonists for preventing the progression of chronic kidney disease. Cochrane Database Syst Rev. 2020 Oct 27;10(10):CD007004. doi: 10.1002/14651858.CD007004.pub4. PMID 33107592
- See also: Click here to find information about studies related to Bayer products conducted in Europe — http://www.clinicaltrialsregister.eu/
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/